CLINICAL TRIAL: NCT06623214
Title: Assessment of the Safety and Effectiveness of a Micro Radiofrequency Skin Treatment Device (nebulyft)
Brief Title: Assessment of the Safety and Effectiveness of a Micro-RF Skin Treatment Device (nebulyft）
Acronym: ASEMRSTD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Rebecca Medical Science and Technology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBTBAP202404 V1.0
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Wrinkle Reduction
Keywords: wrinkle reduction

STUDY DESIGN:
Intervention Model Description: This clinical design adopted the single-group target value method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- treatment (Experimental): receive treatment
  Interventions: Device: nebulyft

INTERVENTIONS:
Device: nebulyft — Micro Radiofrequency Skin Treatment Device(nebulyft)

SUMMARY:
The objective of the study is to evaluate the safety, efficacy and usage compliance of the home-use device nebulyft for self-treatment of wrinkles appearance. The participants do treatment 5 time /week and last 4 weeks. Each treatment takes 16min to complete. Photographs will be taken before treatment and 1 month after the completion of treatment to compare the wrinkle scale.

DETAILED DESCRIPTION:
This is a single-arm prospective study aimed at evaluating the safety and efficacy of nebulyft device treatment of facial areas. Nebulyft device is a low-power, radio frequency device designed to reduce facial wrinkles. 42 subjects will be enrolled in a single clinical site.

The included subjects will use the device at specified areas, including the cheek (for nasolabial fold lines), and outer eye corners (for crow's feet lines). Each side of the nasolabial fold receives 4 minutes of treatment, and each outer eye corner receives 4 minutes of treatment too. The total time for each treatment is 16 minutes. The study consists of at least five wrinkle reduction treatments a week at home for four consecutive weeks. The first treatment session will be conducted under the supervision of the principal investigator (PI), and the remaining sessions will be conducted at home, with remote assistance from the PI when necessary.

A Self-selection and Labeling Comprehension study will be conducted that includes three main questions regarding the intended use of the device, treatment areas, and the possibility of using the device according to the contraindications.

A usability study will be conducted as part of the clinical study. The study was divided into several steps. The PI must observe the test subject to ensure compliance with all the procedures.

In the first visit, the independent treatment for wrinkle reduction was performed under the investigator's observation. Patients were asked to rate the pain level and note any problems/difficulties during the treatments.

The subjects perform treatment at home for 4 continuous weeks and return for photography at the end of the treatment. They will be asked to rate the pain level of the treatment during the visit.

The subjects take final photographs 4 weeks after finishing the treatment and rate the overall satisfaction of the treatment.

ELIGIBILITY:
Inclusion Criteria:

All subjects received oral and electronic consent in accordance with local laws and regulations. Informed consent explains the nature and purpose of the study and the potential risks involved in the study, and emphasizes the voluntary nature of the test, and the subjects can exit the study at any time for any reason. All subjects can ask questions about the research and give sufficient time before signing. All informed consent must be signed before the start of the study.

1. Adult subjects aged 25-65.
2. The subjects should understand the information provided about the investigative nature of the treatment, possible benefits and side effects, and sign the Informed Consent Form, including the permission to use photography.
3. The subjects should be willing to comply with the study procedure and schedule, including the follow-up visits, and will refrain from using any other or similar treatment technologies (i.e., Laser, RF, IR) for the facial condition.
4. The subjects will carry on with their usual diet and exercise and will not have a significant weight change during the study.
5. The subjects are able to read the User Manual in English.
6. The subjects should have II-IV Fitzpatrick wrinkle skin type.
7. The subjects should have visible facial wrinkles.

Exclusion Criteria:

1. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
2. Permanent implant in the treated area such as metal plates and screws, silicone implants or an injected chemical substance.
3. Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles per investigator's discretion.
4. Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases per investigator's discretion.
5. Pregnancy or nursing, as well as 3-6 months post-childbirth.
6. History of bleeding coagulopathies, or prolonged use of anticoagulants (daily aspirin dosing of 81 mg is acceptable).
7. Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medication per investigator's discretion.
8. Subjects with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regime.
9. Poorly controlled endocrine disorders, such as diabetes or thyroid abnormality per investigator's discretion.
10. Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash per investigator's discretion.
11. History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin per investigator's discretion.
12. Any surgery in treatment area within 3 months prior to treatment or before complete healing.
13. Injected fillers in the treatment area in the last 6 months and Botox in the treatment area in the last 3 month.
14. Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
15. As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the subject.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — doesn't limit
Enrollment: 42 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
wrinkle improvement at least one score point of Fitzpatrick wrinkle scale | From enrollment to the end of treatment at 8 weeks
  Three independent board-certified dermatologists assess patient photographs taken at baseline (before treatment initiation) and compare them to those captured one month after completing the home-based treatment using the Fitzpatrick wrinkle scale, which ranges from 1 (least wrinkles) to 9 (most wrinkles). A treatment is considered successful if at least two of the three evaluators observe reduction of at least one score-point in any of the treated areas; otherwise, it is deemed a failure.

SECONDARY OUTCOMES:
subjective wrinkle improvement in wrinkle appearance as measured by satisfactory questionnaires | From enrollment to the end of treatment at 8 weeks
  Subjective wrinkle improvement is assessed based on participants responses to satisfaction questionnaires. There are four questions in total, each rated on a scale of 1 to 4, where 1 indicates very dissatisfied; and 4 indicates very satisfied. The scores from all four questions are summed up, and the total score is used to determine the participants' overall satisfaction with the treatment results.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Shum, MD, Principal Investigator — DSC Laser &amp;amp; Skin Care Center
Locations (1):
- DSC Laser Skin Care Center, San Gabriel, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
the data will be published on paper